CLINICAL TRIAL: NCT01955369
Title: Amyotrophic Lateral Sclerosis Registry Rhineland-Palatinate
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Responsible Party: Principal Investigator, Joachim Wolf, Senior neurologist of the Dept. of Neurology, Klinikum Ludwigshafen
Other Study IDs: 837.253.09
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: incidence; phenotype; mortality
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Amyotrophic lateral sclerosis patients: Patients were included into the registry if they had a new diagnosis of ALS, a minimum age of 18 years and lived in Rhineland-Palatinate for at least 6 months before date of diagnosis. Diagnosis was based upon the revised El Escorial criteria.

SUMMARY:
There is a lack of prospective and population-based epidemiological data on amyotrophic lateral sclerosis in Germany so far. The purpose of this registry is to investigate the incidence, course and phenotypic variety of ALS in Rhineland-Palatinate, a South-West German state of about 4 million inhabitants.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of amyotrophic lateral sclerosis according to revised El Escorial criteria
* minimum of 18 years
* minimum of 6 months of residency in Rhinelnad-Palatinate

Exclusion Criteria:

* patients below 18 years
* ALS patients outside Rhineland-Palatinate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of the state of Rhineland-Palatinate, Germany (4 million inhabitants)
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wolf, Dr, Principal Investigator — Dept. Neurology, Klinikum Ludwigshafen
Locations (1):
- Dept. of Neurology, Klinikum Ludwigshafen, Ludwigshafen, Germany

REFERENCES:
- [Background] Wolf J, Safer A, Wohrle JC, Palm F, Nix WA, Maschke M, Grau AJ. Factors Predicting Survival in ALS Patients--Data from a Population-Based Registry in Rhineland-Palatinate, Germany. Neuroepidemiology. 2015;44(3):149-55. doi: 10.1159/000381625. Epub 2015 Apr 21. PMID 25895515
- [Result] Wolf J, Wohrle JC, Palm F, Nix WA, Maschke M, Safer A, Becher H, Grau AJ. Incidence of amyotrophic lateral sclerosis in Rhineland-Palatinate, Germany. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Jun;15(3-4):269-74. doi: 10.3109/21678421.2014.887733. Epub 2014 Feb 26. PMID 24571628
- [Result] Wolf J, Safer A, Wohrle JC, Palm F, Nix WA, Maschke M, Grau AJ. Variability and prognostic relevance of different phenotypes in amyotrophic lateral sclerosis - data from a population-based registry. J Neurol Sci. 2014 Oct 15;345(1-2):164-7. doi: 10.1016/j.jns.2014.07.033. Epub 2014 Jul 19. PMID 25086855
- [Result] Wolf J, Safer A, Wohrle JC, Palm F, Nix WA, Maschke M, Grau AJ. Factors predicting one-year mortality in amyotrophic lateral sclerosis patients--data from a population-based registry. BMC Neurol. 2014 Oct 4;14:197. doi: 10.1186/s12883-014-0197-9. PMID 25280575
- See also: Amyotrophic lateral sclerosis registry Rhineland-Palatinate — http://www.als-register.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amyotrophic Lateral Sclerosis Patients
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amyotrophic Lateral Sclerosis Patients
Number analyzed (Participants) | 200
Age, Continuous [Mean (Full Range); unit: years] | 65.8 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: death of participating ALS patients independent of the cause of death
Time Frame: an average of 3 years
Measure: Number; unit: participants
Arm/Group | Amyotrophic Lateral Sclerosis Patients
Number analyzed (Participants) | 200
participants | 134

2. Secondary Outcome: Tracheostomy
Description: tracheostomy in ALS patients following respiratory failure
Time Frame: an average of 3 years
Measure: Number; unit: participants
Arm/Group | Amyotrophic Lateral Sclerosis Patients
Number analyzed (Participants) | 200
participants | 10

3. Other Pre Specified Outcome: Gastrostomy
Description: gastrostomy of ALS patients following weight loss and/or swallowing problems with aspiration
Time Frame: an average of 3 years
Measure: Number; unit: participants
Arm/Group | Amyotrophic Lateral Sclerosis Patients
Number analyzed (Participants) | 200
participants | 49

ADVERSE EVENTS:
Arm/Group | Amyotrophic Lateral Sclerosis Patients
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes